CLINICAL TRIAL: NCT04001764
Title: Comparison of the Efficacy of Radial Artery Catheterization in Three Different Regions in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: direnctez
Record Dates: First submitted 2019-06-15; First posted 2019-06-28 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Arterial Cannulation in Intensive Care Unit; Catheterization, Peripheral; Radial Artery
Keywords: Arterial Catheterization; Peripheral Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The first group (Active Comparator): The radial artery catheterization with ultrasound-guided short axis out of plane intervention will be performed over 2 cm of the wrist for this group.
  Interventions: Procedure: The radial artery cannulation over 2 cm of the wrist
- The second group (Experimental): The radial artery catheterization will be performed in the distal 3/4 area of the forearm with ultrasound-guided short axis out of plane intervention.
  Interventions: Procedure: The radial artery cannulation in the distal 3/4 area of the forearm
- The third group (Experimental): The radial artery catheterization will be performed in the distal 1/2 area of the forearm with ultrasound-guided short axis out of plane intervention.
  Interventions: Procedure: The radial artery cannulation in the distal 1/2 area of the forearm

INTERVENTIONS:
Procedure: The radial artery cannulation over 2 cm of the wrist — The radial artery catheterization performed as short axis out-of-plane with USG over 2 cm of the wrist.
  Arms: The first group
Procedure: The radial artery cannulation in the distal 3/4 area of the forearm — The radial artery catheterization will be performed in the distal 3/4 area of the forearm with ultrasound-guided short axis out of plane intervention.
  Arms: The second group
Procedure: The radial artery cannulation in the distal 1/2 area of the forearm — The radial artery catheterization will be performed in the distal 1/2 area of the forearm with ultrasound-guided short axis out of plane intervention.
  Arms: The third group

SUMMARY:
In this prospective, randomized, open-labeled study, the intensive care patients will be selected for ultrasound-guided cannulation of the radial artery in three different regions. Patients will be divided into three groups with simple randomization. The first group will be determined as 'G1' and the radial artery catheterization with ultrasound-guided short axis out of plane intervention will be performed over 2 cm of the wrist for this group. On the second group (G2), radial artery catheterization will be performed in the distal 3/4 area of the forearm with ultrasound-guided short axis out of plane intervention. On the third group (G3), radial arterial catheterization will be performed in the distal 1/2 area of the forearm with ultrasound-guided short axis out of plane interference. Whether there is a difference in the duration of use of arterial cannula, first entry success rates, duration of intervention, number of procedures, the number of cannulas used and the effects on early and late complications and advantages between the groups will be investigated.

DETAILED DESCRIPTION:
In patients requiring frequent arterial blood gas sampling in the intensive care unit and in cases requiring continuous blood pressure monitoring, arterial cannulation is preferred. The use of USG has also become widespread in anesthesia practice. It is supported by studies that USG-guided interventions cause fewer complications compared to classical methods and reduce intervention time. USG-guided arterial catheterization method is based on the principle of direct visualization of the artery and catheter via USG. In this technique, the catheter and the needle tip are displayed simultaneously with the USG guided to the artery lumen. Imaging of anatomical structures with USG has resulted in a reduction of complications and shortening of the processing time. In the USG screen, adjacent anatomical formations such as veins and nerve structures are simultaneously displayed. This reduces the risk of complications.

Two different techniques are used for USG mediated radial artery cannulation. The first one is the in-plane technique, which forms the long axis image of the arteries by positioning the USG probe to parallel to the vein, and the second is the out-of-plane technique, which forms a short axis image with the probe positioned perpendicular to the arteries.

The ideal location of radial artery catheterization with USG or the advantages/disadvantages of the catheterization zone are not available.

In this randomized prospective and open-label study, patients will be divided into three groups. The first group will be determined as 'G1' and the radial artery catheterization with ultrasound-guided short axis out of plane intervention will be performed over 2 cm of the wrist for this group. On the second group (G2), radial artery catheterization will be performed in the distal 3/4 area of the forearm with ultrasound-guided short axis out of plane intervention. On the third group (G3), radial arterial catheterization will be performed in the distal 1/2 area of the forearm with ultrasound-guided short axis out of plane interference. Comparison of these three groups, in terms of duration of use of arterial cannula, initial entry success rates, duration of intervention, number of procedures used, number of cannulas used and effects on early and late complications, and advantages if any is intended.

Patients will be randomly distributed to three groups. Diagnosis, age, sex, height, weight, and body mass index of the patients will be recorded. The random distribution of obese patients to groups will be ensured. Allen test will be done to the patients before the intervention. Radial artery catheterization will be applied only to patients with the collateral flow. Each group will be measured and recorded before, during and after the intervention. Before the intervention, local anesthetic infiltration will be applied and asepsis will be provided. Early complications (such as hematoma, hemorrhage) and late complications (such as circulatory disorders) will be observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Admission of the first degree relatives of the patients and if the patient can give consent
* Patients over 18
* Non-pregnant patients
* Patients without inotropic/vasopressor support
* Patients who do not have contraindications for radial artery cannulation (thrombosis in the distal region, a focus of infection at the site of entry, lack of adequate collateral flow in the Allen test, peripheral vascular diseases [eg, Raynaud's disease)]

Exclusion Criteria:

* Patient/Patient's first degree relatives refuse to work
* Patients under 18
* Pregnant patients
* Patients with contraindications for radial artery cannulation (thrombosis in the distal region, a focus of infection at the site of entry, lack of adequate collateral flow in the Allen test, peripheral vascular diseases [eg, Raynaud's disease)]
* Patient's inotropic/vasopressor support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Duration of Use of Arterial Cannula | During Procedure
  From the time arterial cannula is successfully inserted until cannula cannot use

SECONDARY OUTCOMES:
Initial Entry Success Rates | During procedure
  Success or fail of initial entry
Duration of Intervention | During procedure
  Time from the beginning of procedure and successful cannulation of radial artery
Number of Punctures | During procedure
  Count of punctures until successful artery cannulation
Early Complications | During procedure
  Complications seen during procedure
Late Complications | Up to 7 days
  Complications seen after successful completion of artery cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Zeki T. TEKGUL, Assoc. Prof., Study Director — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

REFERENCES:
- [Background] Hansen MA, Juhl-Olsen P, Thorn S, Frederiksen CA, Sloth E. Ultrasonography-guided radial artery catheterization is superior compared with the traditional palpation technique: a prospective, randomized, blinded, crossover study. Acta Anaesthesiol Scand. 2014 Apr;58(4):446-52. doi: 10.1111/aas.12299. Epub 2014 Mar 3. PMID 24588456
- [Background] Quan Z, Tian M, Chi P, Cao Y, Li X, Peng K. Modified short-axis out-of-plane ultrasound versus conventional long-axis in-plane ultrasound to guide radial artery cannulation: a randomized controlled trial. Anesth Analg. 2014 Jul;119(1):163-169. doi: 10.1213/ANE.0000000000000242. PMID 24806143
- [Background] Levin PD, Sheinin O, Gozal Y. Use of ultrasound guidance in the insertion of radial artery catheters. Crit Care Med. 2003 Feb;31(2):481-4. doi: 10.1097/01.CCM.0000050452.17304.2F. PMID 12576955
- [Background] Shiver S, Blaivas M, Lyon M. A prospective comparison of ultrasound-guided and blindly placed radial arterial catheters. Acad Emerg Med. 2006 Dec;13(12):1275-9. doi: 10.1197/j.aem.2006.07.015. Epub 2006 Nov 1. PMID 17079789
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140